CLINICAL TRIAL: NCT02499224
Title: A Phase I Study to Assess the Safety, Tolerability, and Pharmacokinetics of YYB101, Hepatocyte Growth Factor (HGF)-Neutralizing Humanized Monoclonal Antibody (Mab), in Advanced Solid Tumors Patients Who Are Refractory to Standard Therapy
Brief Title: Safety and Pharmacokinetics Study of YYB101 in Advanced Solid Tumors Patients Who Are Refractory to Standard Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CellabMED (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV110501-101
Record Dates: First submitted 2015-05-14; First posted 2015-07-16 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2016-03

CONDITIONS: Solid Tumors
MeSH Terms: interventions — monoclonal antibody YYB-101

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YYB101 (Experimental): Dose-escalation cohort: YYB101 of each dose level (0.3mg/kg to 5mg/kg), IV infusion on Day 1, Day 29, and followed by every 2 weeks Dose-expansion cohort: YYB101 of MTD (or RP2D), IV infusion every 2 weeks
  Interventions: Drug: YYB101

INTERVENTIONS:
Drug: YYB101 — Dose-escalation cohort: YYB101 of each dose level (0.3mg/kg to 5mg/kg), IV infusion on Day 1, Day 29, and followed by every 2 weeks until disease progression or unacceptable toxicity development.
  Dose-expansion cohort: YYB101 of MTD (or RP2D), IV infusion every 2 weeks until disease progression or unacceptable toxicity development

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and maximum tolerated dose (MTD) of YYB101, HGF-neutralizing humanized Mab, in advanced solid tumors patients who are refractory to standard therapy.

DETAILED DESCRIPTION:
To evaluate the safety, tolerability, and pharmacokinetics of YYB101, patients who are refractory to standard therapy will be enrolled in this study. In dose-escalation cohort, subjects will be enrolled sequentially into four dose cohorts receiving a single dose of YYB101 (0.3, 1, 3, or 5 mg/kg; 3 or 6 subjects per dose cohort) and will be entered the 4-week treatment-free period to evaluate safety and pharmacokinetics. If no dose-limiting toxicity (DLT) is observed during the 4-week period, YYB101 administration will be resumed at the same dose level every 2 weeks until disease progression or unacceptable toxicity development. After the completion of the dose-escalation cohort, additional subjects will be enrolled into a dose-expansion cohort at the maximum tolerated dose (MTD) or recommended phase II dose (RP2D) for further exploration of safety, tolerability, efficacy and pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 19 years or older
2. Patients with pathologically or cytologically confirmed advanced solid tumor which is refractory to standard treatment or for which there is no standard therapy
3. ECOG performance status ≤ 2
4. Life expectancy of ≥ 12 weeks
5. Adequate hematologic, hepatic and renal functions as follows:

   * ANC ≥ 1,500/µL (without G-CSF support within 2 weeks before IP administration)
   * Platelet ≥ 100,000/µL (without transfusion within 2 weeks before IP administration)
   * Hemoglobin ≥ 10.0 g/dL (without transfusion within 4 weeks before IP administration)
   * Serum creatinine ≤ 1.5 mg/dL or eGRF ≥ 60 mL/min/1.73 m2
   * AST and ALT ≤ 2.5 x ULN (AST and ALT ≤ 5 x ULN in the presence of liver metastasis or hepatocarcinoma)
   * Total bilirubin ≤ 1.5 x ULN (with exception of the case associated with Gilbert's syndrome)
   * PT and aPTT ≤ 1.5 x ULN
   * UPC < 1.0 (g/g) (requiring if protein ≥ 1 positive (+) in urinalysis)
6. Patients who voluntarily give written informed consent

Exclusion Criteria:

1. Patients with hematologic malignancies including lymphoma
2. Chemo-, radio-chemo-, biologic-, immuno- or radiotherapy for advanced solid tumor within 4 weeks (or nitrosoureas, mitomycin within 6 weeks or targeted biological antibody within 8 weeks) before IP administration
3. Patients had received high-dose chemotherapy requiring hematopoietic progenitor cell support within 2 years before IP administration
4. Patients with symptomatic central nervous system (CNS) metastasis (patients who are radiologically and neurologically stable condition for ≥ 4 weeks and discontinued corticosteroids at least 4 week before IP administration are able to participate in this trial.)
5. History of deep vein thrombosis or pulmonary embolism within 1 year; Cytomegalovirus (CMV), Epstein-Barr virus (EBV), acute coronary syndrome (including unstable angina or myocardial infarction), or clinically significant cerebrovascular disease (including stroke) within 6 month; Major surgery requiring general anesthesia or respiratory assist within 4 weeks (or video-assisted thoracoscopic surgery or open-and-closed surgery within 2 weeks) before IP administration
6. Concurrent NYHA class III or IV heart failure, uncontrolled hypertension, poorly controlled arrhythmia, other clinically significant cardiovascular abnormalities at investigator's discretion (e.g. LVEF < 50%, clinical significant abnormalities of heart wall, or cardiac muscle damage), known positive result for HIV or other uncontrolled active infection disease
7. Requirement for continuous non-steroidal anti-inflammatory drugs (NSAIDs) or systemic corticosteroids
8. Receiving anticoagulant, history of bleeding diathesis, massive hemoptysis, gastrointestinal hemorrhage, or peptic ulcer disease (< 325 mg aspirin is acceptable)
9. History of severe drug hypersensitivity or hypersensitivity to IP or similar Mab
10. Pregnancy or breast-feeding
11. Women of childbearing potential (WOCBP) or men who are unwilling to use adequate contraception or be abstinent during the trial and for at least 2 months after the end of treatment
12. Patients who received investigational product or investigational device in other clinical trials within 3weeks prior to participation in this trial
13. Patients who cannot participate in this trial at the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Dose-escalation cohort: DLTs and MTD | 28 days

SECONDARY OUTCOMES:
Incidence of AEs that result in discontinuation and dose reduction of YYB101 | By 12 months after enrollment of the last subject
Clinical laboratory abnormalities that result in discontinuation and dose reduction of YYB101 | By 12 months after enrollment of the last subject
Vital sign that result in discontinuation and dose reduction of YYB101 | By 12 months after enrollment of the last subject
Anti-YYB101 antibody that result in discontinuation and dose reduction of YYB101 | By 12 months after enrollment of the last subject
Area under the plasma concentration versus time curve (AUC) of YYB101 | By 4 and 8 weeks after last administration, average 16 weeks
Peak Plasma Concentration (Cmax) of YYB101 | By 4 and 8 weeks after last administration, average 16 weeks

OTHER OUTCOMES:
Serum HGF Concentration profile according to YYB101 dosing | By 12 months after enrollment of the last subject
Tissue cMET expression level before YYB101 dosing | By 12 months after enrollment of the last subject
  Tissue cMET expression level and efficacy (Best overall response, Progress-free survival, Disease control rate)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Jung Yong, MD, Ph.D, Study Director — National OncoVenture/National Cancer Center; Hong SungHee, MS, Study Director — National OncoVenture/National Cancer Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim ST, Hong JY, Park SH, Park JO, Park YW, Park N, Lee H, Hong SH, Lee SJ, Song SW, Kim K, Park YS, Lim HY, Kang WK, Nam DH, Lee JW, Park K, Kim KM, Lee J. First-in-human phase I trial of anti-hepatocyte growth factor antibody (YYB101) in refractory solid tumor patients. Ther Adv Med Oncol. 2020 Jun 2;12:1758835920926796. doi: 10.1177/1758835920926796. eCollection 2020. PMID 32536979